CLINICAL TRIAL: NCT03327649
Title: Neuromodulation of Inflammation to Treat Heart Failure With Preserved Ejection Fraction
Brief Title: Neuromodulation to Treat Patients With Heart Failure With Preserved Ejection Fraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8251
Record Dates: First submitted 2017-10-27; First posted 2017-10-31 (Actual); Results first posted 2022-09-22 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure With Normal Ejection Fraction
Keywords: heart failure with preserved ejection fraction; inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Sham control (Sham Comparator): Patients will receive 1 hour of sham transcutaneous low level vagal stimulation daily for 3 months
  Interventions: Device: low level transcutaneous vagus nerve stimulation
- Active treatment (Experimental): Patients will receive 1 hour of active transcutaneous low level vagal stimulation daily for 3 months
  Interventions: Device: low level transcutaneous vagus nerve stimulation

INTERVENTIONS:
Device: low level transcutaneous vagus nerve stimulation — Stimulation of the auricular branch of the vagus nerve

SUMMARY:
Heart failure with preserved ejection fraction (HFpEF) is a leading cause of mortality in the elderly. Outcomes of patients with HFpEF are poor and so far, no treatment has been shown to decrease morbidity or mortality. Recent animal and human studies suggest that a systemic proinflammatory state, produced by comorbidities, including aging, plays a central role in the development of HFpEF, supporting the notion that attenuating the proinflammatory state is an attractive therapeutic target for HFpEF. We have previously shown that low-level transcutaneous electrical stimulation of the vagus nerve (tVNS) suppresses inflammation in patients with atrial fibrillation. The overall objective of this proposal is to examine the effects of tVNS on diastolic dysfunction, exercise capacity and inflammation in patients with HFpEF. Our specific aims include: 1. To examine the effect of intermittent (1 hour daily for 3 months) tVNS on diastolic dysfunction and exercise capacity, relative to sham stimulation, in patients with HFpEF and 2. To examine the effect of intermittent (1 hour daily for 3 months) LLTS on inflammatory cytokines relative to sham stimulation, in patients with HFpEF. The proposed proof-of-concept studies will provide the basis for the design of further human studies using LLTS among populations with HFpEF. In light of the increasing number of elderly patients with HFpEF and the poor success of the currently available treatment options, an alternative and novel approach such as tVNS has the potential to impact clinical practice and improve health outcomes among a large number of patients. It is anticipated that these investigations will contribute to the broader understanding of the role of inflammation in the pathogenesis of HFpEF and how its inhibition can be used to provide therapeutic effects. Moreover, it is anticipated that a better understanding of how modulation of inflammation affects one of the hallmarks of HFpEF, diastolic dysfunction, will lead to the development of novel pharmacological and non-pharmacological approaches to treat this disease.

ELIGIBILITY:
Inclusion Criteria:

* HFpEF, defined as signs and symptoms of heart failure, LV ejection fraction ≥50%, brain natriuretic peptide ≥35pg/mL and echocardiographic evidence of diastolic dysfunction (left atrial volume index ≥34mL/m2, mitral E-wave velocity/mitral annular velocity ratio [E/e']≥13 and e'<9cm/s) plus 2 of the following 4 comorbidities:

  * age ≥ 65,
  * diabetes,
  * hypertension and
  * obesity, defined as body mass index ≥30kg/m2

Exclusion Criteria:

* LV ejection fraction <40%
* significant valvular disorder (i.e., prosthetic valve or hemodynamically significant valvular diseases)
* recent (<6 months) stroke, myocardial infarction or hospitalization for heart failure
* severe heart failure (class III or IV)
* end stage kidney disease
* recurrent vasovagal syncope
* history of vagotomy
* pregnancy
* sick sinus syndrome and 2nd or 3rd degree AV block (without a pacemaker).

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Stavrakis, MD, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Yes
A biologic repository will be maintained and consideration of its use for future research (linked only to de-identified data) will be integrated into the initial informed consent process for this study. Data needed for independent verification of research results will be made publicly available within 12 months of the end of the funding period (and any no-cost extension).
Time Frame: 12 months after study completion

REFERENCES:
- [Derived] Goggins E, Inoue H, Okusa MD. Neuroimmune Control of Inflammation in Acute Kidney Injury and Multiorgan Dysfunction. J Am Soc Nephrol. 2025 Dec 1;36(12):2473-2484. doi: 10.1681/ASN.0000000813. Epub 2025 Jul 7. PMID 40622772
- [Derived] Stavrakis S, Elkholey K, Morris L, Niewiadomska M, Asad ZUA, Humphrey MB. Neuromodulation of Inflammation to Treat Heart Failure With Preserved Ejection Fraction: A Pilot Randomized Clinical Trial. J Am Heart Assoc. 2022 Feb;11(3):e023582. doi: 10.1161/JAHA.121.023582. Epub 2022 Jan 13. PMID 35023349

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sham Control | Active Treatment
Started | 26 | 26
Completed | 24 | 24
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham Control | Active Treatment | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 15
  >=65 years | 16 | 17 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.3 (9.1) | 69.8 (8.8) | 70.1 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 8 | 8 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 20 | 19 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 24 | 48

OUTCOME MEASURES:

1. Primary Outcome: E/e' (Early Mitral Inflow Doppler Velocity to the Early Diastolic Mitral Annulus Velocity)
Description: E/e' was measured by echocardiography. E/e' correlates very well with left ventricular end diastolic pressure. Higher numbers indicate elevated left ventricular end diastolic pressure.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Sham Control | Active Treatment
Number analyzed (Participants) | 24 | 24
ratio | 10.4 (1.5) | 9.9 (1.5)

2. Primary Outcome: Global Longitudinal Strain
Description: Global longitudinal strain was measured by echocardiography. It is a measure of longitudinal shortening of the myocardium as a percentage (change in length as a proportion to baseline length), thus explaining the negative values. Reduced global longitudinal strain has been associated with adverse clinical outcomes irrespective of left ventricular ejection fraction.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percentage of myocardial shortening
Arm/Group | Sham Control | Active Treatment
Number analyzed (Participants) | 24 | 24
percentage of myocardial shortening | -16.1 (2.5) | -18.6 (2.5)

3. Secondary Outcome: Exercise Capacity
Description: 6 minute walk test
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Sham Control | Active Treatment
Number analyzed (Participants) | 24 | 24
meters | 326.9 (140.4) | 352.7 (158.8)

4. Secondary Outcome: Inflammatory Cytokines
Description: Serum inflammatory cytokines (tumor necrosis factor-alpha)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Sham Control | Active Treatment
Number analyzed (Participants) | 24 | 24
pg/mL | 11.3 (2.5) | 8.7 (2.2)

5. Secondary Outcome: Minnesota Living With Heart Failure Questionnaire
Description: The Minnesota Living with Heart Failure Questionnaire is a well validated measure of quality of life in patients with heart failure. It can have a score 0 to 105, with higher scores reflecting worse quality of life.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham Control | Active Treatment
Number analyzed (Participants) | 24 | 24
units on a scale | 36.6 (14.8) | 23.8 (14.8)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Sham Control | Active Treatment
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 3/24 | 4/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham Control (N=24) | Active Treatment (N=24)
hospitalization (Cardiac disorders) | 3 (3) | 4 (4) — hospitalization for heart failure or persistent atrial fibrillation. Hospitalizations were considered a non-serious adverse event and were not related to the intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-16): https://cdn.clinicaltrials.gov/large-docs/49/NCT03327649/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-10): https://cdn.clinicaltrials.gov/large-docs/49/NCT03327649/ICF_001.pdf